CLINICAL TRIAL: NCT04765800
Title: Differential Efficacy of Guided Imagery Psychotherapy: Comparing Guided Imagery Psychotherapy and Unified Psychodynamic Protocol Therapy for Emotional Disorders in a Non-Inferiority RCT and with Regard to Differential Indication
Brief Title: Differential Efficacy of Guided Imagery Psychotherapy: Non-Inferiority Trial and Exploration of Differential Indication
Acronym: DE-GIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kassel (Other)
Collaborators: Deutsche Gesellschaft für Katathym Imaginative Psychotherapie (DGKIP) (Unknown); International Psychoanalytic University Berlin (Other)
Responsible Party: Principal Investigator, Christian Sell, Principal Investigator, International Psychoanalytic University Berlin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DiW-KIP
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Emotional Disorders
Keywords: depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Non-Inferiority Trial (NI margin: d = 0.46, required N = 152, α = 0.025, 1-β = 0.80)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unified Psychodynamic Protocol for Emotional Disorders (UPP-EMO) (Active Comparator): manualized treatment with a focus on core psychodynamic treatment principles; no use of imagery-based interventions.
  Interventions: Behavioral: weekly, biweekly, or twice a week sessions of face-to-face outpatient psychotherapy
- Guided Imagery Psychotherapy for Emotional Disorders (GIP-EMO) (Experimental): manualized treatment with regular applications (every 4-5 sessions) of guided affective imagery; the therapeutic work is explicitly focused on the patient's guided imagery.
  Interventions: Behavioral: weekly, biweekly, or twice a week sessions of face-to-face outpatient psychotherapy

INTERVENTIONS:
Behavioral: weekly, biweekly, or twice a week sessions of face-to-face outpatient psychotherapy — according to the German Psychotherapy Guidelines (Richtlinie des Gemeinsamen Bundesausschusses über die Durchführung der Psychotherapie)

SUMMARY:
The DE-GIP study compares the efficacy and differential efficacy of two manualized psychodynamic psychotherapies for emotional disorders. The study therefore has two independent aims:

A) The first aim is to test the hypothesized non-inferiority (NI margin: 5 points in PHQ-ADS, requiring N = 152 for a one-sided α = 0.025 and 1-ß = 0.80) of Guided Imagery Psychotherapy for Emotional Disorders (GIP-EMO) to the established Unified Psychodynamic Protocol for Emotional Disorders (UPP-EMO). The primary outcome is anxiety and depression severity (as measured by the PHQ-ADS) 12 months after the beginning of treatment.

B) The second aim is to assess whether GIP-EMO is more effective for patients meeting the GIP suitability criteria (as measured by the Suitability Questionnaire for Guided Imagery Psychotherapy) than for patients who do not meet these criteria. Furthermore, it will be tested whether GIP-EMO is more effective than UPP-EMO for patients who meet the GIP suitability criteria.

DETAILED DESCRIPTION:
Background: Guided Imagery Psychotherapy (GIP) is an established therapeutic method in several countries. In addition to applying the established principles of psychodynamic psychotherapy, the GIP practitioner also regularly conducts sessions in which the patient is asked to imagine their own version of a pre-determined motif (e.g., a mountain or a house) and immediately describe it to the therapist. The patient is meant to allow the image to spontaneously develop further, and to experience its sensual properties while remaining in dialogue with the therapist. The therapist aims to guide and deepen the imagery process by asking questions about the patient's bodily and emotional experiencing and sometimes also by suggesting certain courses of action within the patient's imagined scenery. The patient is instructed to draw his imagery in between sessions. During non-imagery sessions, therapist and patient jointly work to understand the patient's spontaneous imagery within a psychodynamic framework and relate it back to the patient's psychological difficulties. GIP is especially aimed at treating patients with depression, anxiety as well as psychosomatic conditions.

Design and aims: This is a two-arm randomized non-inferiority trial. In addition, the study is used to explore and test possible differential indications of GIP. Manualized GIP for emotional disorders (GIP-EMO) is tested against the manualized psychodynamic therapy according to the unified psychodynamic protocol for emotional disorders (UPP-EMO) as an active comparator. The aim is to test two independent hypotheses: 1) GIP-EMO is non-inferior (NI margin: 5 points in the PHQ-ADS (d = 0.46) requiring N = 152, α = 0.025, 1-ß = 0.80) to UPP-EMO with regard to anxiety and depression severity 12 months after the beginning of treatment. 2) There is a subgroup of patients for whom GIP-EMO is particularly effective. The investigatorshave developed a therapist-questionnaire (Suitability Questionnaire for Guided Imagery Psychotherapy) to assess potential GIP suitability criteria in the patients of the sample. The investigators expect that GIP-EMO is more effective for patients meeting the GIP suitability criteria than for patients who do not meet these criteria. Furthermore, it will be tested whether GIP-EMO is more effective than UPP-EMO for patients who meet the GIP suitability criteria.

Interventions, patient recruitment, and measurements: The interventions in both treatment conditions are regarded as forms of psychodynamic psychotherapy by German legal standards. They are therefore equally eligibly for financial coverage by statutory health insurances. Currently, up to 24 sessions of psychodynamic psychotherapy require only a formal notification to the health insurance. After that, therapist and patient need to file an application for long-term treatment, entailing up to 100 sessions in total. Sessions are in the face-to-face setting and can be weekly, biweekly, or twice a week. The study design does not impose any further requirement regarding treatment length or frequency of sessions. Patients are recruited trough the participating therapists in their private practices. Baseline assessment and eligibility check takes place prior to randomization, that is: after the initial telephone contact between patient and therapist. The assessment includes online questionnaires for the patient and the therapist as well as a SCID interview for the patient. The interviews are conducted via telephone by trained research assistants. For the duration of the treatment, patients complete monthly online questionnaires. After the end of treatment, they complete the same questionnaire every three months. All therapy sessions will be audio-recorded so that treatment fidelity can be assessed by independent raters (Comparative Psychotherapy Process Scale; Process Scale for Imagery- and Trance-Based Psychodynamic Therapies). The primary outcome assessment takes place 12 months after the beginning of treatment and is thus independent of length of treatment or treatment condition. Further follow-up assessments are conducted until 48 months after the beginning of treatment.

Non-inferiority specifications and sample size determination: the investigators determined the margins of non-inferiority (NI) based on the recommendation that the threshold for NI be set to the minimum clinically important difference (MCID) of the primary outcome scale. The MCID was determined as follows: in validation studies for the PHQ-ADS, the authors recommend using either a 1-SEM (standard error of measurement) change (3 to 4 points in the PHQ-ADS) or a 2-SEM change (6 to 8 points in the PHQ-ADS) as MCID. As a compromise, the investigators chose 5 points in the PHQ-ADS as MCID for this study, which is equivalent to an effect size of d = 0.46 given the mean SD of 10.87 found across the three samples of the PHQ-ADS validation study. As a result, the investigators accept the non-inferiority of GIP-EMO to UPP-EMO if the upper limit of the one-sided 0.975 CI of the adjusted mean difference between treatments in favor of UPP-EMO is 5 or below. To test the non-inferiority hypothesis at a one-sided 2.5% significance level with a power of 80%, n = 76 patients are needed per treatment condition. The final sample size includes an oversampling to compensate for an expected loss of 15% to the 12-month follow-up.

Statistical analyses: the investigators shall use intention to treat (ITT) analysis (including all patients who were randomized), using linear-mixed effect models to appropriately deal with repeated measures, nested data, and missing values. Duration and total number of sessions will be included as covariates and therapists as a random coefficient. The investigators shall also use multiple imputations by chained equations to account for data missing at random in the primary outcome. Additional modified ITT analyses (including only patients who started treatment) and per protocol analyses (including only patients who completed treatment) will be conducted to assess the robustness of the results.

ELIGIBILITY:
Inclusion Criteria:

* depressive disorder, anxiety disorder or somatic symptom disorder (with comorbid depressive or anxiety disorder) according to German version of the DSM-5 (SCID-5-CV, Beesdo-Baum et al., 2019) as main diagnosis
* informed consent to participate voluntarily in the study
* sufficient German language skills to understand the patient-report questionnaires

Exclusion Criteria:

* acute suicidality
* diagnosis of schizophrenia, schizophreniform, schizoaffective disorders, and/or psychosis NOS
* bipolar disorder
* depressive disorder with mood-incongruent psychotic features
* paranoid/ schizotypal/ borderline/ or antisocial personality disorder
* severe neurological disorder
* PTSD with intrusive re-experiencing
* clinically relevant substance dependence
* psychopharmacological treatment other than antidepressants
* other simultaneous psychological treatments
* organic cause of depression/anxiety or drug-induced depression/anxiety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety and depression severity as measured by the PHQ-ADS | 12 months after the beginning of treatment
  German version of the Patient Health Questionnaire Anxiety and Depression Scale [range: 0-48]; higher scores indicate more symptom distress through anxiety and/or depression; non-inferiority margin: d = 0.46 = 5 points in the PHQ-ADS (s. NI specifications in the study description)

SECONDARY OUTCOMES:
Somatic symptom severity as measured by the PHQ-15 | 12 and 48 months after the beginning of treatment
  Total somatic symptom severity score of the German version of the Patient Health Questionnaire [range: 0-30]; higher scores indicate more symptom distress through somatic symptoms
Quality of life as measured by the WHOQOL-BREF | 12 and 48 months after the beginning of treatment
  Overall quality of life score of the German version of the WHO Quality of Life-BREF [range: 0-100]; higher scores indicate better quality of life
Severity of interpersonal problems as measured by the IIP-32 | 12 and 48 months after the beginning of treatment
  German version of the Inventory of Interpersonal Problems 32 [range: 0-4]; higher scores indicate more severe interpersonal problems
Levels of personality functioning as measured by the LPFS-BF | 12 and 48 months after the beginning of treatment
  German version of the Level of Personality Functioning Scale-Brief Form [range: 1-4]; higher scores indicate more personality pathology
Levels of Structural integration as measured by the OPD-SQS | 12 and 48 months after the beginning of treatment
  OPD Structure Questionnaire Brief [range: 0-4]; higher scores indicate more personality pathology
Self-efficacy as measured by the module "self-efficacy" from the HEALTH-49 | 12 and 48 months after the beginning of treatment
  Hamburg Modules for the Assessment of Psychosocial Health [range: 0-4]; higher scores indicate less self-perceived efficacy
Difficulties in emotion regulation as measured by the DERS-SF | 12 and 48 months after the beginning of treatment
  Difficulties in Emotion Regulation Scale Short Form [range: 1-5]; higher scores indicate worse emotion regulation
Alexithymia as measured by the TAS-26 | 12 and 48 months after the beginning of treatment
  German version of the Toronto Alexithymia Scale [range: 26-130]; higher scores indicate lower ability to identify and describe emotions
Utilization of Medical Services and Work Incapacity Periods | 12 and 48 months after the beginning of treatment
  German version of the Questionnaire for the Assessment of the Utilization of Medical Services as well as Work Incapacity Periods; higher scores indicate higher associated health care costs and/or more work incapacity days
Clinically meaningful overall improvement as measured by the CGI-I | 12 months after the beginning of treatment
  Therapist-rating of the Clinical Global Impression - Improvement [range: 1-7]; improvement is indicated by scores < 4

CONTACTS AND LOCATIONS:
Overall Officials: Christian Sell, Prof., Principal Investigator — International Psychoanalytic University Berlin; Cord Benecke, Prof., Principal Investigator — University of Kassel
Locations (1):
- University of Kassel, Kassel, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler M, Petersen G, Vu HM, Baudry M, Lynch G. L-phenylalanyl-L-glutamate-stimulated, chloride-dependent glutamate binding represents glutamate sequestration mediated by an exchange system. J Neurochem. 1987 Apr;48(4):1191-200. doi: 10.1111/j.1471-4159.1987.tb05646.x. PMID 2880930
- [Background] Sell C, Schöpfer-Mader E, Brömmel B & Möller H (2017). Therapeutisches Vorgehen und Interventionen in Katathym Imaginativer Psychotherapie, Hypnosepsychotherapie und Autogener Psychotherapie: Entwicklung und Validierung der Therapeutenversion der 'Prozessskala für imaginations- und trancebasierte tiefenpsychologische Methoden' (PIT). Psychotherapie Forum, 22(4), 113-126. https://doi.org/10.1007/s00729-017-0102-2
- [Background] Hilsenroth MJ, Blagys MD, Ackerman SJ, Bonge DR & Blais MA (2005). Measuring Psychodynamic-Interpersonal and Cognitive-Behavioral Techniques: Development of the Comparative Psychotherapy Process Scale. Psychotherapy: Theory, Research, Practice, Training, 42(3), 340-356. https://doi.org/10.1037/0033-3204.42.3.340
- [Background] Kroenke K, Wu J, Yu Z, Bair MJ, Kean J, Stump T, Monahan PO. Patient Health Questionnaire Anxiety and Depression Scale: Initial Validation in Three Clinical Trials. Psychosom Med. 2016 Jul-Aug;78(6):716-27. doi: 10.1097/PSY.0000000000000322. PMID 27187854
- [Background] Leichsenring F, Steinert C. Towards an evidence-based unified psychodynamic protocol for emotional disorders. J Affect Disord. 2018 May;232:400-416. doi: 10.1016/j.jad.2017.11.036. Epub 2017 Nov 11. PMID 29522960
- [Background] Gräfe K, Zipfel S, Herzog W, Löwe B (2004): Screening psychischer Störungen mit dem "Gesundheitsfragebogen für Patienten (PHQ-D)." Ergebnisse der deutschen Validierungsstudie. Diagnostica 50, 171-181.
- [Background] Thomas A, Brähler E, Strauß B (2011): IIP-32: Entwicklung, Validierung und Normierung einer Kurzform des Inventars zur Erfassung interpersonaler Probleme. Diagnostica 57, 68-83.
- [Background] Ehrenthal JC, Dinger U, Schauenburg H, Horsch L, Dahlbender RW, Gierk B. [Development of a 12-item version of the OPD-Structure Questionnaire (OPD-SQS)]. Z Psychosom Med Psychother. 2015;61(3):262-74. doi: 10.13109/zptm.2015.61.3.262. German. PMID 26388057
- [Background] Spitzer C, Muller S, Kerber A, Hutsebaut J, Brahler E, Zimmermann J. [The German Version of the Level of Personality Functioning Scale-Brief Form 2.0 (LPFS-BF): Latent Structure, Convergent Validity and Norm Values in the General Population]. Psychother Psychosom Med Psychol. 2021 Jul;71(7):284-293. doi: 10.1055/a-1343-2396. Epub 2021 Mar 10. German. PMID 33694153
- [Background] Rabung S, Harfst T, Kawski S, Koch U, Wittchen HU, Schulz H. [Psychometric analysis of a short form of the "Hamburg Modules for the Assessment of Psychosocial Health" (HEALTH-49)]. Z Psychosom Med Psychother. 2009;55(2):162-79. doi: 10.13109/zptm.2009.55.2.162. German. PMID 19402020
- [Background] Gratz KL, Roemer L (2004). Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. J Psychopathol Behav Assess 26, 41-54. https://doi.org/10.1023/B:JOBA.0000007455.08539.94
- [Background] Kupfer J, Brosig B, Brahler E. [Testing and validation of the 26-Item Toronto Alexithymia Scale in a representative population sample]. Z Psychosom Med Psychother. 2000;46(4):368-384. doi: 10.13109/zptm.2000.46.4.368. German. PMID 11793322
- [Background] Roick C, Kilian R, Matschinger H, Bernert S, Mory C, Angermeyer MC. [German adaptation of the client sociodemographic and service receipt inventory - an instrument for the cost of mental health care]. Psychiatr Prax. 2001 Oct;28 Suppl 2:S84-90. doi: 10.1055/s-2001-17790. German. PMID 11605129
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Beesdo-Baum K, Zaudig M, Wittchen H-U (2019). SCID-5-CV: Strukturiertes Klinisches Interview für DSM-5-Störungen - Klinische Version. Hogrefe.
- [Background] Leichsenring F, Luyten P, Hilsenroth MJ, Abbass A, Barber JP, Keefe JR, Leweke F, Rabung S, Steinert C. Psychodynamic therapy meets evidence-based medicine: a systematic review using updated criteria. Lancet Psychiatry. 2015 Jul;2(7):648-60. doi: 10.1016/S2215-0366(15)00155-8. Epub 2015 Jun 30. PMID 26303562
- [Background] Friedrichs-Dachale A, Ullmann H (2020): Katathym Imaginative Psychotherapie (KIP). Eine systematisch aufgebaute, vielseitig anwendbare Methode der psychodynamischen Psychotherapie. Psychodynamische Psychotherapie 2/2020, 153-173. DOI 10.21706/pdp-19-2-153
- [Background] Lesaffre E. Superiority, equivalence, and non-inferiority trials. Bull NYU Hosp Jt Dis. 2008;66(2):150-4. PMID 18537788